# **COVER PAGE**

| Study protocol | |
|----------------|----------------------------------|
| Title | Safety and Performance of the |
| | Motorized Spiral Endoscope |
| | (PowerSpiral) in Subjects |
| | indicated for small-bowel |
| | enteroscopy or Endoscopic |
| | Retrograde Cholangio- |
| | Pancreatography (ERCP) in |
| | Subjects with surgically altered |
| | gastrointestinal anatomy: |
| | A PMCF Registry |
| Short Title or | The SAMISEN study |
| Acronym | (SAfety and Performance of |
| | the MotorIzed Spiral |
| | ENdoscope) |
| NCTNumber | NCT05129449 |



# SCLINICAL INVESTIGATION PLAN

Safety and Performance of the
Motorized Spiral Endoscope
(PowerSpiral) in Subjects indicated
for small-bowel enteroscopy or
Endoscopic Retrograde CholangioPancreatography (ERCP) in Subjects
with surgically altered
gastrointestinal anatomy:
A PMCF Registry

SAfety and Performance of the MotorIzed Spiral
Endoscope - The SAMISEN study

**Investigational Device:** 



**Sponsor:** Olympus Europa SE & Co. KG

Motorized Spiral Endoscope (PowerSpiral) INTESTINAL

VIDEOSCOPE OLYMPUS PSF-1 in combination with SINGLE

USE POWERSPIRAL TUBE DPST-1 used with the motor control

unit POWERSPIRAL CONTROL UNIT PSCU.

**CIP Reference No.:** 2018-GI (OEKG) – 01

**Document Version:** Final Version 03

Elaboration Date: 28-Jun-2021

Amendments: 02



THE STUDY WILL BE CONDUCTED IN COMPLIANCE WITH THE DECLARATION OF HELSINKI, GOOD CLINICAL PRACTICE (GCP), DIN (EN) ISO 14155:2020, AND ALL APPLICABLE NATIONAL LAWS AND REGULATIONS.

### **Confidential Information**

This clinical investigation plan is the confidential information of Olympus Europa SE & Co. KG and is intended solely for guidance of the clinical investigation. This investigation plan may not be disclosed to parties not associated with this clinical investigation or used for any purpose without the prior written consent of Olympus Europa SE & Co. KG.

CIP Reference No.:2018-GI (OEKG) -01. The **SAMISEN** study - Final Version 03 - Date 28-Jun-2021

# SIGNATURE PAGE

| Manager | Clinical | Operations: |
|---------|----------|-------------|
|---------|----------|-------------|

Name, Title: Peter Teichmann, PhD

Institution: Olympus Europa SE & Co. KG

Street: Wendenstraße 20 Zip code - City: 20097 Hamburg

Country: Germany

Hamburg, 28-Jun-2021

Date Signature

**Coordinating Clinical Investigator:** 

Name, Title: Torsten Beyna, MD PhD

Professional Position: Senior Consultant and Head of Gastroenterology Unit

Department of Internal Medicine

Institution: Evangelisches Krankenhaus Düsseldorf

Street: Kirchfeldstraße 40
Zip code – City: 40217 Düsseldorf

Country: Germany

Sept 10 2021

Date

Confidential


# Co-Coordinating Clinical Investigator:

Name, Title:

Tom Gustaaf Moreels, Prof MD PhD

Professional Position:

Division of Gastroenterology & Hepatology

Institution:

Cliniques universitaires Saint-Luc

Street:

Hippokrateslaan 10

Zip code - City:

B-1200 Brussels

Country:

Belgium

Date

Brumb 30 AV4 221

## Statistician

Name, Title

Carsten Schwenke, PhD

Institution

SCO:SSiS

Street

Karmeliterweg 42

Zip code City

13465 Berlin

Country

Germany

Berlin, 13/AUG/2021

Date

Signature


# **DECLARATION OF PRINCIPAL INVESTIGATOR**

I have read this clinical investigation plan (CIP) and agree that it contains all the information required to conduct the trial. I agree to conduct the trial as set out in this CIP. I will not enroll the first subject in the trial until I have received approval for conduct of this study from the appropriate ethics committee and until all legal requirements have been fulfilled. I agree to obtain in the manner described in the CIP a written informed consent to participate from all subjects enrolled in this study and to keep the dated and signed consent forms for 15 years.

| Site number: | < Enter Site number here> |
|-------------------------|---------------------------|
| Principal Investigator: | < Enter name of PI here> |
| Place, Date | Signature Investigator |


# **CONTACT ADDRESSES AND RESPONSIBILITIES**

Manager Clinical Operations Peter Teichmann, PhD

Olympus Europa SE & Co. KG

Wendenstraße 20

20097 Hamburg, Germany

Email: peter.teichmann@olympus-europa.com

Phone: +49 40 23773 7835 Fax: +49 40 23773 507835

Coordinating Clinical Investigator

Torsten Beyna, MD PhD

Evangelisches Krankenhaus Düsseldorf

Kirchfeldstraße 40

40217 Düsseldorf, Germany

Co-Coordinating Clinical Investigator

Tom G. Moreels, MD PhD

Cliniques universitaires Saint-Luc

Hippokrateslaan 10

B-1200 Brussels, Belgium

**Safety Contact** 

Peter Teichmann, PhD

Olympus Europa SE & Co. KG

Wendenstraße 20

20097 Hamburg, Germany

Email: peter.teichmann@olympus-europa.com

Phone: +49 40 23773 7835 Fax: +49 40 23773 507835

**CRO** 

Eberhard Buchner, PhD

Winicker Norimed GmbH Medizinische Forschung

Samisen study team Deutschherrnstraße 15-19

90429 Nürnberg, Germany


# Statistician

Carsten Schwenke, PhD SCO:SSiS Karmeliterweg 42 13465 Berlin, Germany


# **TABLE OF CONTENTS**

| Signature | Page | 4 |
|---|---|---|
| Declaration | on of Principal Investigator | 6 |
| Contact A | ddresses and Responsibilities | 7 |
| Table of ( | Contents | 9 |
| List of abl | previations and definitions | . 13 |
| Trial Sum | mary | . 14 |
| 1 Bac | kground and Rationale | . 17 |
| 1.1 D | escription of the Investigational Device | . 18 |
| 1.2 J | ustification for the Design of the Clinical Investigation | . 18 |
| 1.3 R | isks and Benefits | . 20 |
| 2 Tria | l Objectives | . 22 |
| 2.1 C | bjective | . 22 |
| 3 Des | ign of the Clinical Investigation | . 23 |
| 3.1 G | eneral | . 23 |
| 3.1.1 | Design Overview | . 23 |
| 3.1.2 | Randomization and Blinding or Assignment of Investigational Device | . 23 |
| 3.1.3 | Variables in the Clinical Investigation | . 23 |
| 3.1.4 | Replacement of Subjects | . 24 |
| 3.2 lr | vestigational Device(s) and Comparators | . 24 |
| 3.2.1 | Investigational Device(s) | . 24 |
| 3.2.2 | Comparator Devices(s) | . 24 |
| 3.2.3 | Reference Device(s) | . 24 |
| 3.2.4 | Other Medical Device / Medication | . 24 |
| 3.3 S | ubjects | . 24 |
| 3.3.1 | Inclusion criteria | . 24 |
| 3.3.2 | Exclusion criteria | . 26 |
| 3.3.3 | Subject Withdrawal or discontinuation | . 26 |
| 3.3.4 | Point of Enrolment | . 26 |
| 3.3.5 | Duration of the Clinical Investigation | . 27 |


| | 3.3 | .6 | Sample size | 27 |
|---|---|---|---|---|
| 3 | 3.4 | Pr | ocedures | 28 |
| | 3.4 | .1 | Overview of the Procedures and Laboratory Measurements | 28 |
| | 3.4 | .2 | Description of clinical investigation related procedures and assessed data | 28 |
| | 3.4 | .3 | Study Visits Schedule | 32 |
| | 3.4 | .4 | Concomitant treatments | 32 |
| | 3.4 | .5 | Medical Care after Termination of the Clinical Investigation | 33 |
| | 3.4 | .6 | Deviations from medical standard | 33 |
| 3 | 3.5 | M | onitoring Plan | 33 |
| | 3.5 | .1 | Responsibilities | 33 |
| | 3.5 | .2 | Source Data Definition and Verification (SDV) | 33 |
| 4 | 5 | Stati | sticis | 35 |
| 4 | 1.1 | St | atistical methods | 35 |
| | 4.1 | .1 | Background and demographic characteristics | 35 |
| | 4.1 | .2 | Efficacy evaluation | 35 |
| | 4.1 | .3 | Safety evaluation | 36 |
| | 4.1 | .4 | Interim analysis | 36 |
| | 4.1 | .5 | Other evaluations | 36 |
| 4 | 1.2 | Sı | ıbgroup Analyses | 36 |
| 4 | 1.3 | Mi | ssing/spurious Data | 37 |
| 5 | I | Data | Management | 38 |
| 5 | 5.1 | Da | ata recording | 38 |
| 5 | 5.2 | Da | ata processing | 38 |
| 6 | , | Ame | ndments to the CIP | 39 |
| 7 | ( | CIP I | Deviations | 40 |
| 8 | | Devi | ce Accountability | 41 |
| 9 | 9 | State | ment of Compliance | 42 |
| ç | 9.1 | Et | hical and Regulatory Aspects | 42 |
| ç | 9.2 | Pa | atient Coverage | 42 |
| ç | 9.3 | Re | etention of Documents | 42 |


| 9.4 A | Auditing procedures | 43 |
|---|---|---|
| 10 Info | rmed Consent | 44 |
| 11 Adv | verse Events, Adverse Device Effects and DevIce Deficiencies | 45 |
| 11.1 | Definitions (according to ISO 14155:2020) | 45 |
| 11.1.1 | Adverse event (AE) | 45 |
| 11.1.2 | Adverse Device Effect (ADE) | 45 |
| 11.1.3 | Serious Adverse Event / Serious Adverse Device Effect (SAE /SADE) | 46 |
| 11.1.4 | Device Deficiencies | 47 |
| 11.2 | Documentation | 47 |
| 11.2.1 | (Serious) Adverse Events / Adverse Device Effects | 47 |
| 11.2.2 | Device deficiencies | 48 |
| 11.3 F | Reporting Responsibilities | 48 |
| 11.3.1 | Serious Adverse Events (SAE) / Serious Adverse Device Effects (SADE) | 48 |
| 11.3.2 | Device deficiencies | 48 |
| 11.3.3 | Responsible Nominated Safety Contact | 48 |
| 11.4 A | Anticipated Adverse Events | 49 |
| 11.5 | Data Monitoring Committee | 51 |
| 12 Vuli | nerable Population | . 52 |
| 13 Sus | pension or Premature Termination | 53 |
| 14 Pub | olication Policy | . 54 |
| 15 Bibl | liography | . 55 |
| 16 Stud | dy Timeline | . 57 |
| 17 Ann | nex 01: Deep Enteroscopy PROCEDURE | . 58 |
| 17.1 | General Information | . 58 |
| 17.2 | General Insertion tips | . 58 |
| 17.3 | General Withdrawal tips | . 58 |
| 17.4 A | Antegrade Approach | . 59 |
| 17.4.1 | Inserting the Scope | . 59 |
| 17.4.2 | Passing through the Pharynx & Esophagus | . 60 |
| 17.4.3 | Passing through the Stomach | 61 |

| | CIP Reference No.:2018-GI (OEKG) -01. The <b>SAMISEN</b> study - Final Version 03 - Date 28-Jun-2021 |
|---|---|
| 17.4.4 | Passing through the Duodenum |
| 17.4.5 | Passing through the Small Bowel Distal to the Ligament of Treitz |
| 17.4.6 | Reaching the Terminal Ileum64 |
| 17.4.7 | Withdrawal Techniques65 |
| 17.5 R | etrograde Approach |
| 17.5.1 | Passing through the Colon |
| 17.5.2 | Eliminating a Loop |
| 17.5.3 | Passing through the Ileo-cecal Valve |
| 17.5.4 | Passing through the Small Bowel |
| 17.5.5 | Reaching the Proximal Jejunum71 |
| 17.5.6 | Withdrawal Techniques72 |
| Table of t | ables |
| Table 2 L | st of study procedures |


# LIST OF ABBREVIATIONS AND DEFINITIONS

| Abbreviation | Definition |
|--------------|------------------------------------------------------------|
| ADE | Adverse Device Effect |
| AE | Adverse Event |
| ATC | Anatomical Therapeutic Chemical |
| BAE | Balloon assisted enteroscopy |
| CE | Commission Européen |
| CIP | Clinical Investigation Plan |
| CCI | Coordinating Clinical Investigator |
| CRF | Case Report Form |
| CRO | Contract Research Organization |
| CV | Curriculum vitae |
| DBE | Double balloon enteroscopy |
| DIMDI | German Institute for medical documentation and information |
| EC | Ethics Committee |
| ECG | Electrocardiogram |
| ERCP | Endoscopic Retrograde Cholangiopancreatography |
| GCP | Good Clinical Practice |
| ICH | International Conference on Harmonization |
| ISF | Investigator Site File |
| PI | Principal Investigator |
| PTC | Percutaneous transhepatic cholangiography |
| SADE | Serious Adverse Device Effect |
| SAE | Serious Adverse Event |
| SBE | Single balloon enteroscopy |
| SOP | Standard Operating Procedure |
| SDV | Source Data Verification |
| TMF | Trial Master File |
| U | Unit |
| WHO | World Health Organization |


# **TRIAL SUMMARY**

| Title | Safety and Performance of the Motorized Spiral Endoscope (PowerSpiral) in Subjects indicated for small-bowel enteroscopy or Endoscopic Retrograde Cholangio-Pancreatography (ERCP) in Subjects with surgically altered gastrointestinal anatomy: A PMCF Registry |
|---|---|
| Short Title or<br>Acronym | The SAMISEN study (SAfety and Performance of the MotorIzed Spiral ENdoscope) |
| Version/<br>Date | CIP#: 2018-GI (OEKG) – 01<br>Version 3.0 (28-Jun-2021)<br>PHASE B: ERCP in patients with surgically altered GI anatomy (Roux-en-Y and Billroth II types). |
| Sponsor | OLYMPUS EUROPA SE & Co. KG<br>Amsinckstraße 63<br>20097 Hamburg, Germany |
| Purpose | Demonstrate safety and clinical performance of the Motorized Spiral Endoscope (PowerSpiral) in daily medical practice. |
| Objective | Prospectively collect clinical data on the application of the Motorized Spiral Endoscope (PowerSpiral) in a typical clinical setting within the Intended Use. |
| Endpoints | Parameter for analysis: |
| | <ul> <li>Total success rate: Defined as the combined percentage of Enteroscopy<br/>success rate, Biliary Cannulation success rate and Procedural<br/>(Therapeutic) success rate.</li> </ul> |
| | <ul> <li>Enteroscopy success rate: Defined as the percentage of procedures<br/>with the ability to reach the major papilla or the biliary anastomosis.</li> </ul> |
| | <ul> <li>Biliary Cannulation success rate: Defined as the percentage of<br/>procedures with the ability to selectively cannulate the bile duct and<br/>conduct a cholangiography.</li> </ul> |
| | <ul> <li>Therapeutic (Procedural) success rate: Defined as the percentage of<br/>procedures in which the intended treatment could be successfully<br/>completed.</li> </ul> |
| | <ul> <li>Total procedure time: (starting with oral insertion until final withdrawal of<br/>the device).</li> </ul> |
| | <ul> <li>Enteroscopy time: (starting with oral insertion until reaching the papilla or the biliary anastomosis).</li> </ul> |
| | <ul> <li>Safety: Incidence (% of subjects) and frequency (no. of subjects) with<br/>Serious Adverse Events (SAEs) and Device Deficiencies (DD) which<br/>meet the severity grading of moderate or severe for the following<br/>categories:</li> </ul> |
| | <ul> <li>Enteroscopy-associated complications (mainly bleeding and perforation(s))</li> <li>ERCP-related complications (Dumonceau et al. 2020)</li> <li>Sedation / anesthesia related complications</li> <li>other</li> </ul> |
| | User feedback and assessment of handling characteristics of the device. |
| Study Design | International, multicenter, open label, non-randomized, prospective, observational study. |
| Sample Size | The study consists of two phases: Phase A which comprises deep enteroscopies only [completed by the time Phase B will start] and Phase B, |


| For Phase B: Approximately 4-5 sites experienced both in conventional ERCP as well as in ERCP in patients presenting with previous GI surgery will proceed to Phase B of this study. 00 (ERCP) patients will be enrolled in this exploratory study. Study Start (Enrollment of First Patient) is planned for Phase B in November 1021. Enrollment period: approximately 12-18 months. Study closure of Phase B is expected before end of 2022. Please note: Phase B will start after completion of Phase A. The results from the Phase A will be reported independently from Phase B. Motorized Spiral Endoscope (PowerSpiral) INTESTINAL VIDEOSCOPE DLYMPUS PSF-1 in combination with SINGLE USE POWERSPIRAL TUBE DPST-1 used with the motor control unit POWERSPIRAL CONTROL UNIT PSCU. Subjects presenting with surgically altered GI anatomy indicated for ERCP with biliary indication, which fulfil all inclusion and none of the exclusion riteria: Inclusion criteria Signed informed consent |
|---|
| ERCP as well as in ERCP in patients presenting with previous GI surgery will proceed to Phase B of this study. 00 (ERCP) patients will be enrolled in this exploratory study. Study Start (Enrollment of First Patient) is planned for Phase B in November 1021. Enrollment period: approximately 12-18 months. Study closure of Phase B is expected before end of 2022. Please note: Phase B will start after completion of Phase A. The results from the Phase A will be reported independently from Phase B. Motorized Spiral Endoscope (PowerSpiral) INTESTINAL VIDEOSCOPE DLYMPUS PSF-1 in combination with SINGLE USE POWERSPIRAL TUBE DPST-1 used with the motor control unit POWERSPIRAL CONTROL UNIT PSCU. Subjects presenting with surgically altered GI anatomy indicated for ERCP with biliary indication, which fulfil all inclusion and none of the exclusion riteria: Inclusion criteria Signed informed consent |
| Enrollment period: approximately 12-18 months. Study closure of Phase B is expected before end of 2022. Please note: Phase B will start after completion of Phase A. The results from the Phase A will be reported independently from Phase B. Motorized Spiral Endoscope (PowerSpiral) INTESTINAL VIDEOSCOPE DLYMPUS PSF-1 in combination with SINGLE USE POWERSPIRAL TUBE DPST-1 used with the motor control unit POWERSPIRAL CONTROL UNIT PSCU. Subjects presenting with surgically altered GI anatomy indicated for ERCP with biliary indication, which fulfil all inclusion and none of the exclusion criteria: Inclusion criteria Signed informed consent |
| Enrollment period: approximately 12-18 months. Study closure of Phase B is expected before end of 2022. Please note: Phase B will start after completion of Phase A. The results from the Phase A will be reported independently from Phase B. Motorized Spiral Endoscope (PowerSpiral) INTESTINAL VIDEOSCOPE DLYMPUS PSF-1 in combination with SINGLE USE POWERSPIRAL TUBE DPST-1 used with the motor control unit POWERSPIRAL CONTROL UNIT PSCU. Subjects presenting with surgically altered GI anatomy indicated for ERCP with biliary indication, which fulfil all inclusion and none of the exclusion criteria: Inclusion criteria Signed informed consent |
| Please note: Phase B will start after completion of Phase A. The results from the Phase A will be reported independently from Phase B. Motorized Spiral Endoscope (PowerSpiral) INTESTINAL VIDEOSCOPE DLYMPUS PSF-1 in combination with SINGLE USE POWERSPIRAL TUBE DPST-1 used with the motor control unit POWERSPIRAL CONTROL UNIT PSCU. Subjects presenting with surgically altered GI anatomy indicated for ERCP with biliary indication, which fulfil all inclusion and none of the exclusion criteria: Inclusion criteria Signed informed consent |
| Please note: Phase B will start after completion of Phase A. The results from the Phase A will be reported independently from Phase B. Motorized Spiral Endoscope (PowerSpiral) INTESTINAL VIDEOSCOPE DLYMPUS PSF-1 in combination with SINGLE USE POWERSPIRAL TUBE DPST-1 used with the motor control unit POWERSPIRAL CONTROL UNIT PSCU. Subjects presenting with surgically altered GI anatomy indicated for ERCP with biliary indication, which fulfil all inclusion and none of the exclusion criteria: Inclusion criteria Signed informed consent |
| Phase A will be reported independently from Phase B. Motorized Spiral Endoscope (PowerSpiral) INTESTINAL VIDEOSCOPE DLYMPUS PSF-1 in combination with SINGLE USE POWERSPIRAL TUBE DPST-1 used with the motor control unit POWERSPIRAL CONTROL UNIT PSCU. Subjects presenting with surgically altered GI anatomy indicated for ERCP with biliary indication, which fulfil all inclusion and none of the exclusion writeria: Inclusion criteria Signed informed consent |
| DLYMPUS PSF-1 in combination with SINGLE USE POWERSPIRAL TUBE DPST-1 used with the motor control unit POWERSPIRAL CONTROL UNIT PSCU. Subjects presenting with surgically altered GI anatomy indicated for ERCP with biliary indication, which fulfil all inclusion and none of the exclusion writeria: Inclusion criteria Signed informed consent |
| OPST-1 used with the motor control unit POWERSPIRAL CONTROL UNIT PSCU. Subjects presenting with surgically altered GI anatomy indicated for ERCP with biliary indication, which fulfil all inclusion and none of the exclusion writeria: Inclusion criteria Signed informed consent |
| vith biliary indication, which fulfil all inclusion and none of the exclusion riteria: nclusion criteria . Signed informed consent |
| nclusion criteria . Signed informed consent |
| . Signed informed consent |
| Detients with surgically altered upper Contraintentinal anotomy (Doug on V |
| Patients with surgically altered upper Gastrointestinal anatomy (Roux-en-Y and Billroth II types) with a biliary indication for ERCP where access with conventional ERCP devices is of no avail and after careful risk assessment. |
| xclusion criteria |
| n addition to be eligible for study enrollment a subject must not meet any of he exclusion criteria listed below. |
| <ol> <li>Age under 18 years</li> <li>Female and of child-bearing age who is currently pregnant or planning to become pregnant within the study period</li> <li>Any contraindication to standard enteroscopy or ERCP (e.g. severe coagulopathy or known coagulation disorder; bowel obstruction / stenosis, stents or other instruments implanted in the intestinal tract, suspected GI perforation, esophageal or gastric varices, eosinophilic esophagitis) as judged by the investigator after careful individual risk assessment</li> <li>Concurrent participation in another competing clinical study</li> <li>Pancreatic indication for ERCP in patient with surgically altered anatomy</li> </ol> |
| Each subject will undergo the following study visits: |
| <ul> <li>Visit 1 – screening visit, inform potential subjects about the trial, obtain informed consent from subjects to participate in the study, check inclusion / exclusion criteria, collect data on medical history and concomitant medication.</li> <li>Visit 2 - scheduled procedure: perform ERCP as planned. Provide feedback on the handling characteristics of the PowerSpiral enteroscope.</li> <li>[Visit 3 - Only for Phase A, not applicable anymore for Phase B (an optional) second procedure: retrograde (or antegrade) enteroscopy as necessary.]</li> <li>Visit 4 - pre-hospital discharge visit: collect any (delayed) complication the study team will monitor observed SAEs on a regular (daily, but at least weekly)</li> </ul> |
| n he |


| Study Flow<br>Chart | Patient selection | Visit 1 | Visit 2 | Visit 3 – (optional for<br>Phase A.<br>NA for Phase B) | Visit 4 |
|---|---|---|---|---|---|
| | | Screening visit | Scheduled procedure | Second scheduled procedure | Hospital discharge visit |
| | Patient scheduled for enteroscopy of small-bowel no | Inclusion / yesexclusion criteria | Anterograde and/or retrograde enteroscopy or ERCP as planned | Anterograde or retrograde enteroscopy if necessary | → Final visit |
| Study<br>Contacts | Sponsor: OLYMPUS EUROPA SE & Co. KG Wendenstraße 20 20097 Hamburg, Germany Manager Clinical Operations: Peter Teichmann, PhD Manager Clinical Operations email: peter.teichmann@olympus- europa.com phone: +49 40 23773 7835 mobile: +49 170 5570 674 Coord. Clin. Investigator (CCI): Torsten Beyna, MD PhD Dept. of Internal Medicine Ev. Krankenhaus Düsseldorf Kirchfeldstraße 40 40217 Düsseldorf, Germany Co-CCI Prof. Tom Gustaaf Moreels, MD P Cliniques universitaires Saint-Luc Division of Gastroenterology & He Hippokrateslaan 10 B-1200 Brussels, Belgium | | rf<br>y<br>, MD PhD<br>nt-Luc | | |


# 1 BACKGROUND AND RATIONALE

Small bowel enteroscopy is usually performed in order to evaluate gastrointestinal bleeding, small bowel tumors, polyps, inflammatory or other small bowel diseases. Video capsule endoscopy, single- (SBE), double-balloon (DBE) or spiral enteroscopy are the most popular non-surgical endoscopic techniques in this context. Hereof the endoscopic approach offers additional diagnostic and therapeutic options as biopsies and direct therapeutic intervention is possible compared to capsule endoscopy. These enteroscopy systems – also called overtube-assisted enteroscopy (OAE) techniques - are used to visualize the small-bowel and proceed with a therapeutic intervention, either during the same or in a subsequent session. For example, the DBE utilizes distal and proximal balloons that can be inflated and deflated to "anchor" and move the bowel, thereby assisting the operator in advancing the endoscope while gathering the bowel onto the overtube shaft.

However, the SBE and DBE procedures are time consuming and usually require 2 operators to perform this kind of examination.

Patients with altered upper gastrointestinal (upper GI) anatomy (such as Roux-en-Y gastric bypass) indicated for Endoscopic Retrograde Cholangio-Pancreatography (ERCP) represent a special challenge to the investigator and require a well-experienced endoscopist (Krutsri et al. 2019). With the growing acceptance of bariatric surgery the number of patients requiring ERCP has significantly increased (Anvari et al. 2021). Current state of the art is performing ERCP with single/double balloon devices. Limited data with the manual spiral device ERCP promising results have been obtained so far (Lennon et al. 2012).

It is generally considered as a safe procedure with a low risk of serious adverse events (Moreels 2019). Complication rates with SBE/DBE or rotational overtube enterscopy devices in this patient population were reported in the range of 4% up to 12% (Skinner et al. 2014). In an actual systematic review article and meta-analysis with 1523 patients the AE rate was just 4 % (Anvari et al. 2021), however Shah et al reported in 129 patients with ERCPs using single-balloon, double-balloon and rotational manual overtube an AE rate of 12,4% (Shah et al. 2013).

The new endoscopic techniques originally designed for deep enteroscopy have increased the potential to reach the area of interest and successfully perform an ERCP and therapeutic interventions with an acceptable complication rate. There were already ERCPs conducted with PowerSpiral as it is within the intended use. Beyna et al. recently published their first clinical case after Roux-en-Y reconstructive surgery and bilioenteric anastomosis was described (Beyna, Schneider, et al. 2020).


# 1.1 Description of the Investigational Device

The Motorized Spiral Enteroscope (INTESTINAL VIDEOSCOPE OLYMPUS PSF-1 and SINGLE USE POWERSPIRAL TUBE DPST-1) in conjunction with the motor control unit (POWERSPIRAL CONTROL UNIT PSCU) now offers a new technology which combines the advantageous options of enteroscopy with a faster and less invasive approach. The intended use of this CE-certified medical device (PowerSpiral) is to examine the lumen of the small intestine to provide clear images for diagnostic and therapeutic purposes in the management and treatment of small-bowel disease.

The system is similar to other currently marketed endoscopes and incorporates a flexible insertion tube, light source, digital imaging, and channels for passing accessories for sample collection or therapeutic interventions. In contrast to the predecessor a novel user-controlled motor rotates a special spiral cuff (SINGLE USE POWERSPIRAL TUBE DPST-1) located on the endoscope's insertion tube (POWERSPIRAL CONTROL UNIT PSCU). Rotation of this cuff, which has soft spiral-shaped "fins", pleats the small bowel on to the endoscope's insertion tube, thereby allowing rapid and atraumatic access into deeper regions of the small bowel. The Rotating speed is 30 rpm and the Rotation torque is controlled mechanically until torque limit is reached (until a limiting function is activated).

With this new medical device system deep enteroscopy allows complete visualization of the small bowel. The motorized PowerSpiral can be used for either antegrade or retrograde approach according to the operator's preference or individual patient anatomy. The new device shall contribute to easier and faster disease clarification and necessary therapeutic interventions in all areas of the small intestine including patients with altered anatomy, e.g. after bariatric surgeries. Also for special procedures like ERCP the PowerSpiral medical device system can be used very well (Beyna, Schneider, et al. 2020; M Schneider 2020) and thus represents an alternative approach to more risky surgical interventions.

The study investigators shall have considerable experience in deep enteroscopy and ERCP. The study team will undergo special training (arranged by the Sponsor) to become comfortable with all handling characteristics of this novel device. The product and procedure training is mandatory prior to enrolling the first study subject and will be documented accordingly.

# 1.2 Justification for the Design of the Clinical Investigation

Deep enteroscopy is well established with Balloon assisted enteroscopy procedures, however there is a need for innovative and faster methods, less resource utilization which at the same time provide more comfort for the patients.

Currently available and published data for PowerSpiral was collected by means of Investigator Initiated Trials (Mans et al. 2018); (Neuhaus et al. 2016); (Beyna, Arvanitakis, Schneider, Gerges, Boing, et al. 2020); (Beyna, Arvanitakis, Schneider, Gerges, Hoellerich, et al. 2020). With this


Olympus sponsored Registry further data about performance and safety for this new medical device will be collected in a larger patient population. Obtained safety data will be compared to data published in respective guidelines or literature.

This study will be performed in parallel to the European market launch of this new medical device. It is a registry study with a CE marked medical device whose application within the intended use will be captured. The registry does not impose any additional procedure or risk beyond standard of care as we strive to document daily clinical routine. Therefor this study is <u>observational</u> (non-interventional) in nature.

For the same reason inclusion criteria are kept as broad as possible. In summary all patients are eligible where the physician realizes an indication for deep enteroscopy in Phase A and Endoscopic Retrograde Cholangio-Pancreatography (ERCP) in Phase B for further diagnostic or therapeutic work up. The exclusion criteria will only affect patients under the age of 18 years and pregnant women. Otherwise clinical judgement of the treating physician is the only relevant and leading reason for exclusion. Of course, giving signed informed consent by all study subjects is a prerequisite for participation in this "registry".

The SAMISEN study consists of two phases (Phase A and B). In the first Phase A the patients receive a deep enteroscopy. In Phase B patients with altered upper GI anatomy indicated for ERCP will be enrolled to investigate clinical safety and performance of PowerSpiral in this special patient cohort.

Patients indicated for ERCP who present with altered upper GI anatomy, e.g. Roux-en-Y, use of PowerSpiral is in line with the intended use as defined by the manufacturer. In all cases, the treating physician will take the final decision after careful assessment of the individual risk.

At the end, the SAMISEN study and analysis will contain data collected for PowerSpiral in the complete area of the intended use. This means deep enteroscopy (Phase A) and ERCP (Phase B). Due to Olympus internal and time reasons the data will be collected consecutively.

For the study Phase A 10 European sites were recruited that offer deep enteroscopy to their patients. For Phase B only 4-5 sites of them will proceed and conduct the ERCP examinations. This <u>international multi-center</u> setup will give a more representative picture and avoid a single-site bias. Furthermore, enrollment will be completed earlier compared to a single center approach.

The prevailing complications of a deep enteroscopy are pancreatitis, perforation, bleeding and adverse events associated with sedation or anesthesia (Aktas et al. 2010; Akarsu et al. 2014; Akerman and Cantero 2009; Arulanandan et al. 2016; He et al. 2013; Moeschler and Mueller 2015). Generally these are independent if the procedure was performed as a diagnostic or therapeutic procedure however the complications rate is usually higher in interventional cases (Rondonotti et al. 2018).

The main objective of the SAMISEN study Phase A was to assess the performance and safety of diagnostic and therapeutic procedures with the newly designed Olympus Motorized Spiral Enteroscope (INTESTINAL VIDEOSCOPE OLYMPUS PSF-1 and SINGLE USE POWERSPIRAL TUBE DPST-1) system in combination with the motor control unit (POWERSPIRAL CONTROL


UNIT PSCU). All Serious Adverse Events (SAE) observed in this study will be documented so the overall SAE rate as well as the number of individual types of complications (bleeding, pancreatitis etc.) can be calculated.

The publication of Rondonotti (Rondonotti et al. 2018) for device-assisted enteroscopy for diagnosis and treatment of small-bowel disorders represents an excellent source for comparison. Hence this study is designed as a <u>prospective study</u> without control group. The resulting SAE rate will be compared to the historical data from this ESGE Technical Review (Rondonotti et al. 2018). The clinical performance will be characterized by calculating the Diagnostic and Therapeutic Yield, Total Procedure Time, time needed for Therapeutic Intervention, Total Small Bowel Enteroscopy Rate and user feedback on device handling.

In Phase B patients will be enrolled to further investigate the efficacy and safety profile in patients with altered upper GI anatomy with an indication for an ERCP examination, as PowerSpiral is a real alternative to reach the bile duct especially in this kind of patient population where a normal duodenoscopy is insufficient for this purpose. Aim of this explorative study setting is to collect efficacy and safety data for an ERCP procedure conducted with PowerSpiral, as there are currently limited clinical data available (Beyna, Schneider, et al. 2020; M Schneider 2020). The study team will monitor the safety reports on a regular basis and SAEs will be evaluated by an independent expert/safety monitor.

### 1.3 Risks and Benefits

Patients with altered upper gastrointestinal anatomy requiring Endoscopic Retrograde Cholangio-Pancreatography (ERCP) represent a special challenge to the endoscopist. Independent of the clinical study this kind of examination has certain clinical risks associated with such a procedure which must be balanced against other treatment alternatives (e.g. open surgery). After careful consideration of risk and benefits the investigator may decide to proceed with direct visualization of the small bowel or perform ERCP to the biliary ductal system. Especially in patients with surgically altered upper gastrointestinal anatomy PowerSpirals offers a new and good option to reach the target area for ERCP, the major papilla or the hepaticojejunal anastomosis to conduct a cholangiopancreatography (Beyna, Schneider, et al. 2020). Due to the non-interventional character of this study (i.e. registry) no additional protocol driven procedures besides medical standard are required. In summary the potential risk(s) a study subject will potentially face is considered identical to the risks he/she would be facing without participating in this study.

The complication rate associated with endoscopic procedures is usually low. Experience with deep enteroscopy of the small-bowel has been published for SBE and DBE. Distribution and incidence of complications depend whether it was a diagnostic or therapeutic approach. For therapeutic procedures tissue usually is removed or biopsies obtained which carries a higher complication rate compared to purely diagnostic procedures. A deep enteroscopy examination is performed with


sedation or anesthesia, depending on the hospital standards. Any anesthesia carries a certain risk for the patient, especially if multi-morbidity is present.

Section 11.4 provides a list of all potential (S)AEs that have either been observed during or after deep enteroscopy or ERCPs with PowerSpiral conducted in a clinical study setting and from the regular usage of this medical device PowerSpiral within the intended use in the field.. There is no additional device related new risk identified that was not already anticipated for its predecessor.

However, the range and incidence of adverse events (AEs) related to endoscopic retrograde cholangiopancreatography (ERCP) differ substantially from those related to other endoscopic procedures. The incidence of the major AEs (pancreatitis, cholangitis, cholecystitis, bleeding, perforation are between 0.08 to 9.7%, Sedation-related AEs up to 24.6% (Dumonceau et al. 2020). As there are currently less safety data for ERCP conducted with PowerSpiral available (Beyna, Schneider, et al. 2020; M Schneider 2020), the study team is committed to check the safety data in detail and regularly to realize at an early stage whether the safety data for PowerSpiral deviates from the frequencies described above. An independent (non recruiting) expert in this field will be involved in the assessment of each SAE captured during Phase B.

The overall risk / benefit ratio for this clinical investigation is assumed to be in the same acceptable range of established balloon assisted methods of deep enteroscopy and enteroscopies conducted for an ERCP examination. PowerSpiral is used regularly in hospitals over the world and every patient has the chance to get an examination with PowerSpiral independent of this study. As mentioned earlier this registry does not impose any additional "protocol driven" interventions or examinations therefore the procedural risk to which a patient will be exposed to should be very similar to the risk in case he/she would not have agreed to participate in this study.


# **2 TRIAL OBJECTIVES**

# 2.1 Objective

The main objective of this registry is to collect data on the safety and performance of the new motorized PowerSpiral device when used as intended by the manufacturer. It is assumed that the new device and its safety profile is non-inferior to preceding generations of balloon assisted enteroscopes.

As clinical performance and efficacy is equally important for the user this study also collects efficacy and handling data of the new device.

With this study OLYMPUS complies with Post-Market Clinical Follow-up (PMCF) requirements.


# 3 DESIGN OF THE CLINICAL INVESTIGATION

#### 3.1 General

### 3.1.1 Design Overview

SAMISEN is an international, multicenter, non-randomized, prospective, observational open label study examining the CE- marked PowerSpiral (OLYMPUS PSF-1, SINGLE USE POWER SPIRAL TUBE and motor control unit POWER SPIRAL CONTROL) device. (For justification of the study design please refer to section 1.2). Phase B has an explorative study design for data collection in ERCP conducted with PowerSpiral.

### 3.1.2 Randomization and Blinding or Assignment of Investigational Device

SAMISEN is designed as a prospective single-arm trial without control group or randomization. All subjects enrolled will undergo one procedure with the Motorized Spiral Endoscope (PowerSpiral).

### 3.1.3 Variables in the Clinical Investigation

It is a prospective and observational Registry without any additional procedure beyond clinical practice. The small-bowel enteroscopy for Phase A and ERCP for Phase B has to be performed according the medical standard. Serious Adverse Events (SAE) and Device Deficiencies (DD) must be documented.

For phase B the following parameters will be analyzed:

- Total success rate: Defined as the combined percentage of Enteroscopy success rate,
   Biliary Cannulation success rate and Procedural (Therapeutic) success rate.
- Enteroscopy success rate: Defined as the percentage of procedures with the ability to reach the major papilla or the biliary anastomosis.
- Biliary Cannulation success rate: Defined as the percentage of procedures with the ability to selectively cannulate the bile duct and conduct a cholangiography.
- Therapeutic (Procedural) success rate: Defined as the percentage of procedures in which the intended treatment could be successfully completed.
- Total procedure time: (starting with oral insertion until final withdrawal of the device).
- Enteroscopy time: (starting with oral insertion until reaching the papilla or the biliary anastomosis).
- Safety: Incidence (% of subjects) and frequency (no. of subjects) with Serious Adverse
  Events (SAEs) and Device Deficiencies (DD) which meet the severity grading of
  moderate or severe for the following categories:
  - Enteroscopy-associated complications (mainly bleeding and perforation(s))

| CIP | Reference No.:2018-GI (OEKG) -01. The <b>SAMISEN</b> study - Final Version 03 - Date 28-Jun-2021 |
|---|---|
| | ERCP-related complications (Dumonceau et al. 2020): |
| | Sedation / anesthesia related complications |
| | other |

User feedback and assessment of handling characteristics of the device.

# 3.1.4 Replacement of Subjects

If subjects enrolled into this study withdraw their consent or drop out for other reasons <u>before</u> the ERCP was actually performed the site shall continue to enroll subjects until the quota of 25 (up to a maximum of 40 patients per individual sites has been reached. Besides that, it is not foreseen to replace subjects that drop out after the first enteroscopy but before hospital discharge.

# 3.2 Investigational Device(s) and Comparators

# 3.2.1 Investigational Device(s)

In this prospective study all investigators will deploy a motorized PowerSpiral device. There are no different (sub)types of this devices, so all devices used will be identical.

#### 3.2.2 Comparator Devices(s)

Not applicable.

#### 3.2.3 Reference Device(s)

Balloon assisted enteroscopy (BAE) devices used for deep enteroscopy and as described in the literature (Rondonotti et al. 2018) will serve as historical controls for Phase A. For Phase B Balloon enteroscopy assisted ERCPs and data from a manual spiral system will be used as reference to compare the phase B results.

#### 3.2.4 Other Medical Device / Medication

Not applicable.

## 3.3 Subjects

#### 3.3.1 Inclusion criteria

In order to be for being eligible for participation in this study subjects presenting with surgically altered GI anatomy indicated for ERCP with biliary indication must meet all of the inclusion criteria listed below to be enrolled into the Phase B of the SAMISEN study:


- Signed informed consent
- Patients with surgically altered upper Gastrointestinal anatomy (Roux-en-Y and Billroth II types) with a biliary indication for ERCP where access with conventional ERCP devices is of no avail and after careful risk assessment



Figure 01: Common types of surgically altered anatomy (Picture from Prof. Tom G. Moreels)


#### 3.3.2 Exclusion criteria

In addition to be eligible for study enrollment a subject must **not** meet any of the exclusion criteria listed below:

- Age under 18 years
- Female and of child-bearing age who is currently pregnant or planning to become pregnant within the study period
- Any contraindication to standard enteroscopy (e.g. severe coagulopathy or known coagulation disorder; bowel obstruction / stenosis, stents or other instruments implanted in the intestinal tract, suspected GI perforation, esophageal or gastric varices, eosinophilic esophagitis) as judged by the investigator after careful individual risk assessment
- Concurrent participation in another competing clinical study
- Pancreatic indication for ERCP in patient with surgically altered anatomy

### 3.3.3 Subject Withdrawal or discontinuation

A subject may withdraw his/her consent to participation at any time without explanation and without consequences for further treatment. Moreover, the study participation may be discontinued temporarily or permanently due to one of the following reasons:

- Any health deterioration of the subject, e.g. ALAT and/or ASAT > 3 times upper limit of normal range,
- 2. Not acceptable further study participation as determined by the investigator,
- 3. Occurrence of not tolerable adverse events and/or laboratory value alterations,
- Technical reasons (change of physician, change of address of subject),
- 5. Lacking compliance of subject,
- Pregnancy,
- 7. Major CIP deviation,
- Subject lost to follow-up,
- 9. Death.

If a subject discontinues participation in the study after signing the consent for whatever reason, every effort has to be made to perform an early termination visit in case the ERCP was already conducted. In this case, the same examinations as in the final visit (Visit 4) shall be performed.

#### 3.3.4 Point of Enrolment

Point of enrolment is defined as the time at which a subject dates and signs the informed consent. At least one day prior to that, the investigator shall provide a complete explanation of the study (benefits, risks, rights and obligations).


# 3.3.5 Duration of the Clinical Investigation

The average duration of study participation for subjects completing the study is estimated to be approximately 2 days up to one week. The estimated total study duration for the whole study cohort is approximately one year. The end of study is defined as the date of the database lock.

## 3.3.6 Sample size

A total of 100 subjects shall be enrolled into SAMISEN study Phase B. As described in section 3.1.1 the study has an explorative design. The sample size was chosen with regards to clinical reasoning with respect to the primary parameter and not on statistical power considerations.

The enrolment period starts in approximately July 2021 and will stop once the expected number of patients per site is reached. This "Last-Patient-In" (end of recruitment) is expected in July 2022.

Each site with two investigators shall take every effort to enroll a balanced number of patients per investigator.

Statistical Analyses will be performed with SAS software version 9.4 (SAS Institute Inc., Cary, NC, USA).


#### 3.4 Procedures

## 3.4.1 Overview of the Procedures and Laboratory Measurements

Table 2 gives an overview of the relevant study procedures:

Table 1 List of study procedures

| Visit | V1 | V2 | V3 | V4 |
|---|---|---|---|---|
| | Screening | 1 <sup>st</sup> scheduled<br>procedure | Optional<br>for Phase A.<br>NA for Phase<br>B | Hospital<br>discharge<br>visit |
| Patient informed consent | х | | | |
| Inclusion/Exclusion criteria | x | | | |
| Demographic data | x | | | |
| Physical examination with vital signs, body measurements (body weight and body height) and concomitant diseases | x | | | |
| Small-bowel<br>enteroscopy / ERCP<br>with PowerSpiral | | x | | |
| Evaluation of criteria regarding usage of PowerSpiral | | x | | |
| (Serious) Adverse<br>Events | | х | | х |

# 3.4.2 Description of clinical investigation related procedures and assessed data

At the screening visit the investigator informs the patient about the trial and selects the patient as potentially suitable for this trial. The patient should receive the patient information and patient consent sheet for information. An official Visit 1 will be arranged.

The following data will be collected during the clinical investigation at the various study visits:

#### At visit V1:

At this visit the patient will be informed about the trial in detail and the patient consent must be signed at Visit 1 (or earlier). All questions of the patient shall be answered.


The following data shall be captured for all patients meeting the inclusion and exclusion criteria:

- Demographic Data
  - Age
  - Sex
- Physical Examination
  - Height
  - Weight
  - Radial pulse (with the subject in the supine position for at least 5 minutes before).
  - Blood pressure (according to Riva Rocci using calibrated sphygmomanometers, the subject has to be in a sitting position for at least 5 minutes, blood pressure will be measured twice within 5 minutes, the mean of both measurements will be calculated).
  - Document if a 12-lead ECG was recorded as medical standard in your hospital.
  - Document if a clinical standard panel of laboratory parameters is determined prior to small-intestine enteroscopy as medical standard in your hospital. Any deviation of laboratory parameters exceeding normal ranges shall be documented and followed up, as appropriate. Clinically significant deviations observed during the screening visit and throughout the study will be documented in the Case Report Form.
  - Select the appropriate ASA class¹ to assess the fitness of the patient.
  - Document any abnormalities detected in one of the following organ systems:
    - Head, neck and thyroid (gland)
    - Skin and mucosa
    - Cardiovascular system
    - Respiratory system
    - Abdomen
    - Spine
    - Extremities
    - Reflexes
    - Other
- Provide information about the following concomitant medication
  - Acetylsalicylic acid

<sup>&</sup>lt;sup>1</sup> We recommend to take the ASA class from the anesthesiologic pre-medication records


- Anticoagulant therapy
- Discontinuation of Anticoagulant therapy prior / during the procedure
- Provide information about previous diagnostic workup:
  - MRCP
  - > CT
  - Sonography
  - > PTC
  - > (Other) Clinical findings without previous imaging
- Details about the biliary indication for ERCP:
  - Suspicious finding from previous diagnostic work up
  - Suspected diagnosis
  - Other
- Planned therapeutic strategy after reaching the papilla or the biliary anastomosis:
  - Stricture treatment
  - Stone treatment
  - Other

# At visit V2

- At this visit the PowerSpiral enteroscopy for ERCP will be performed.
- Enter the date and name of the responsible investigator who performs the enteroscopy.
- Enter the total procedure time ("scope-in, scope-out") measured from initial enteroscope introduction through the bite block to final enteroscope withdrawal through the bite block (minutes) for antegrade approach).
- Provide information about the kind of staff and number persons needed for this enteroscopy.
- Select if a general anesthesia or sedation is used.
- Record total radiation dose (μGy\*m²)
- Answer if the findings of the previous imaging examinations were confirmed or not.
- Please list all therapeutic intervention(s) actually performed:
  - Stent placement
    - Plastic stent


- Metallic stent
- Number of stents
- Stent removal
- Stone extraction
- Intraductal lithotripsy
- Biliary duct dilation
- Biliary sphincterotomy
- Precut sphincterotomy
- Biliary sphincteroplasty
- Dilation of anastomotic stricture
- Biopsy
- Other
- Please indicate if the intervention was successful or not.
- Enter the time needed for any therapeutic intervention. If several slots for therapeutic interventions occurred, please add the time needed for each therapeutic slot and enter the total duration in minutes.
- Answer if any Serious Adverse Events observed during the enteroscopy procedure.
- Document the final diagnosis after the ERCP
- Answer the following questions:
  - Was the therapeutic intervention successful and were all planned therapeutic aim(s) achieved?
  - Was the initial therapeutic management plan modified during the procedure?

After visit 2 the investigator shall give an evaluation of the PowerSpiral procedure in comparison to BAE medical devices for ERCP previously used. The investigator shall judge if the PowerSpiral is "worse", "similar" or "better" than previous equipment used for the following topics:

- Handling (Handling means the whole handling of the instrument (PowerSpiral scope + overtube + motor control unit) during preparation of the equipment and throughout the examination).
- Instrument insertion (Instrument insertion means how the instrument could be inserted.
- Precision of positioning during therapy (This means how precise and how stable the instrument could be positioned during a therapeutic intervention).


- **Time needed for procedure** (It means the time duration describes the start as entering the endoscope in the mouth until withdrawal which suppose as stop point).
- Staff and resources required for procedure.

#### At visit 4

Visit 4 is the hospital discharge visit. The patient is ready to leave the hospital and the status shall be documented.

The following data will be documented:

- Date of the hospital discharge examination.
- Actual discharge date.
- if the patient has recovered from the examination.
- Describe new (Serious) Adverse Event if any
- Clinical signs or symptoms of pancreatitis e.g. elevated Lipase/Amylase (if measured postprocedure as medical standard in your hospital).
- Specify if the patient get further treatment from the referral physician or if additional specialist(s) will be involved.

The investigator will ensure that the patient receives further medication as necessary and can be discharged from hospital and consigned to GP's or medical specialist's care.

Finally, the investigator shall to sign off the eCRF to confirm that the data is complete and accurate.

# 3.4.3 Study Visits Schedule

The standard preparation procedure in your hospital for ERCP shall be followed as usual.

The ERCP duration depends on the individual diagnostic and treatment activities for each patient.

The final visit V4 shall be completed prior to hospital discharge.

Premature study discontinuation of a study subject is to be noted as such on the case report form (eCRF).

### 3.4.4 Concomitant treatments

Concomitant treatment during study participation should be in line with the medical standard for ERCP. Information about Acetylsalicylic acid and Anticoagulant therapy must be documented in the eCRF.


### 3.4.5 Medical Care after Termination of the Clinical Investigation

At the final visit V4 the investigator will ensure that the patient can be discharged from hospital without any identifiable risk and that further treatment on an outpatient basis through a general practitioner or medical specialist will be provided as necessary. Any ongoing (serious) adverse events that deserve special attention shall be mentioned in the patient's discharge letter.

#### 3.4.6 Deviations from medical standard

The observational character of this registry study does not require any additional clinical procedure or tests beyond standard of care. Any deviation for medical reasons shall be documented in the eCRF.

# 3.5 Monitoring Plan

### 3.5.1 Responsibilities

Study monitoring will be performed by the CRO Winicker Norimed GmbH Medizinische Forschung, Nuremberg, Germany and partly the sponsor.

The monitor will visit the study sites in order to check that eCRFs are completed without omission, and that Good Clinical Practice guidelines and the CIP are followed. He/she will also check the progress of subject inclusion. The monitor shall be granted access to the study binder and hospital records of enrolled subjects. The study nurse shall be available to the monitor during monitoring visit(s). The investigator is expected to be available at least for a debriefing at the end of the monitoring site visit.

After study end the site will receive a copy of the eCRF file and the investigator has to ensure that it is stored safely with all other study documents filed in the Investigator Site File according to national law.

# 3.5.2 Source Data Definition and Verification (SDV)

Source data are the original records of all variables collected for the clinical investigation. They include, but are not limited to:

- Signed informed consent,
- Laboratory reports,
- Individual subject clinical notes,
- Hospital charts or pharmacy records and any other similar reports and records of any procedure performed in accordance with the CIP,
- Details concerning inclusion and exclusion criteria.

The investigator must allow the monitor access to all documents in the medical file to confirm their consistency with the electronic case report form entries. All information entered in the eCRF must be available as source data. No information about subject identity on these documents will be


allowed to leave the study site. At a minimum the following points will be verified by the monitor: existence of signed informed consent, adherence to inclusion/exclusion criteria, all SAEs and a tabulation of adverse events. Further checks may be carried out according to the study specific monitoring plan to confirm matching of all eCRF data matches source data.

For more details on Monitoring of this Clinical Investigation please refer to the "Monitoring Plan" (available upon request).


# 4 STATISTICIS

Statistical analysis of the data will be performed by Dr. Carsten Schwenke, SCO:SSiS. The evaluation will be specified in the Statistical Analysis Plan (SAP) laid down in a separate document.

Demographic data, baseline characteristics and information of the physical examination and medical history with concomitant medication will be reported in summary tables. Additional information about the planned procedure covering all endpoints listed below (4.1.2, 4.1.3) will be reported.

# 4.1 Statistical methods

### 4.1.1 Background and demographic characteristics

Continuous variables such as age will be presented by mean, standard deviation, minimum, median and maximum. Categorical data such as gender will be presented as absolute and relative frequencies.

All variables with no coding available will be listed.

# 4.1.2 Efficacy evaluation

The efficacy parameter are defined as follows:

- Total success rate: Defined as the combined percentage of Enteroscopy success rate,
   Biliary Cannulation success rate and Procedural (Therapeutic) success rate.
- Enteroscopy success rate: Defined as the percentage of procedures with the ability to reach the major papilla or the biliary anastomosis.
- Biliary Cannulation success rate: Defined as the percentage of procedures with the ability to selectively cannulate the bile duct and conduct a cholangiography.
- Therapeutic (Procedural) success rate: Defined as the percentage of procedures in which the intended treatment could be successfully completed.
- Total procedure time: (starting with oral insertion until final withdrawal of the device).
- Enteroscopy time: (starting with oral insertion until reaching the papilla or the biliary anastomosis).
- User feedback and assessment of handling characteristics and other logistical aspects regarding:
  - Handling of PowerSpiral
  - Instrument insertion of PowerSpiral

- Precision of positioning during therapy of PowerSpiral
- > Time needed for procedure of PowerSpiral
- Staff and resource needed for procedure of PowerSpiral

No hypothesis testing will be performed for any efficacy endpoint.

## 4.1.3 Safety evaluation

The following safety variables will be collected:

- Enteroscopy-associated Serious adverse events during and after enteroscopy procedure
- ERCP-related Serious adverse events (Dumonceau et al. 2020)
- Sedation / anesthesia related Serious adverse events
- Other Serious adverse events (procedure or product related)
- · Adverse events during enteroscopy and ERCP procedure
- Adverse event of interest are: bleeding, mucosal damage and pancreatitis (including hyperamylasemia)

The safety variables will be tabulated for all study participants.

Adverse events data will be processed in the statistical analysis after coding with the most recent version of MedDRA.

AEs and device deficiencies will be presented in summary tables. These tables will show the number of subjects per group presenting an adverse event and the incidence of its occurrence. Adverse events will be grouped by system organ class and stratified by severity (mild, moderate, severe) and by relation to study treatment (unrelated or related according to the categories definite, probable and possible).

#### 4.1.4 Interim analysis

Not planned.

## 4.1.5 Other evaluations

Not planned.

## 4.2 Subgroup Analyses

Subgroup analysis will be performed on the following subgroups:

- By type of indication (Stone treatment / Stricture treatment)
- By type of reconstructive surgery (BII / Roux-en-Y)
- > By presence / absence of biliodigestive anastomosis (reimplanted papilla)
- First 10 cases vs subsequent cases (to account for learning curve)


# 4.3 Missing/spurious Data

All available data will be included in the analyses and will be summarized as far as possible. Unless otherwise specified there will be no substitution of missing data, i.e. missing data will not be replaced, missing data will be handled as 'missing' in the statistical evaluation.


## 5 DATA MANAGEMENT

## 5.1 Data recording

Data shall be recorded in the eCRFs in a timely manner but not later than 5 working days after collection of the data, including signatures. Please take into account, a SAE must be documented immediately to meet the reporting requirements. The investigator must document all visits and assessments on the respective eCRF form and shall ensure that no empty data blocks exist. If a test or assessment was not performed, the investigator shall indicate this. If a question does not apply, the investigator shall also document this (e.g. by entering "NA").

The investigator shall sign the overall affirmation statement for each patient to document personal responsibility for accuracy, completeness of data captured in the system and for the trial being carried out according to the protocol and any amendments.

Data can only be entered by authorized and trained site staff, i.e. by the investigator or investigator's staff trained on eCRF procedures. (S)AE pages must be signed off by the investigator.

Data corrections in the eCRF done by the investigator or designee require entering a reason for the data change. The change of already entered data and the person who performed the data change will be tracked in the audit trail of the eCRF. In case of data changes in the eCRF that has already been signed off a new signature is required to authorize the data modification.

Queries issued within the eCRF shall be answered within 7 working days.

### 5.2 Data processing

Data processing, controls of plausibility and query handling will be carried out by the CRO Winicker Norimed GmbH Medizinische Forschung, Germany. The study database will be created according to the format and content of the eCRF and the CIP. The MedDRA or IMDRF code will be used for coding of adverse events and previous / concomitant diseases.


## 6 AMENDMENTS TO THE CIP

CIP amendments or supplements (apart from minor administrative changes) require a written amendment. Amendments must be approved by the EC and the regulatory authorities, if locally applicable, before implementation. A copy of the written approvals will be provided to the investigators.

In the following sections are changes compare to CIP version no. 02 from 23th April 2019:

- Contact addresses and responsibilities
- Trial summary
- Section 1
- Section 3.1.1-3.1.4.
- Section 3.2.1
- Section 3.2.3.
- Section 3.3.
- Section 3.3.1.
- Section 3.3.2.
- Section 3.3.3.
- Section 3.3.5.
- Section 3.3.6.
- Section 3.4.1. -3.4.4.
- Section 4.1.2.
- Section 4.1.3.
- Section 4.2.
- Section 5.2.
- Section 6
- Section 8
- Section 11.2.1.
- Section 11.3.3.
- Section 11.4.
- Section 15

Overall, the ISO version was adapted to ISO14155:2020.


## 7 CIP DEVIATIONS

The investigator must not deviate from the procedures described in this CIP.

Under emergency circumstances, deviations from the CIP to protect the rights, safety and well-being of human subjects may proceed without prior approval of the sponsor and the EC. Such deviations must be documented and reported to the sponsor and the EC as soon as possible.

Classifications into minor and major CIP deviations will be performed by the clinical operations manager and statistician at the end of the study.

Major CIP deviations are, but are not restricted to

Deviation from the in- and exclusion criteria


# 8 DEVICE ACCOUNTABILITY

This study is a post-market study. The PS enteroscopes are CE-marked. Hence from a regulatory perspective strict device accountability is not needed. However, the sponsor will have a list of serial numbers and can track which device was delivered to which study site.

The devices are usually purchased by the site. Olympus will provide devices as loaner equipment to a limited number of sites serving as centers of excellence. Any loaner equipment shall be exclusively used for the examination of study patients. After reaching the agreed quota per site (approximately 25 patients, see also 3.1.4) the device must be returned to Olympus. Details are specified in the Clinical Trial Agreements.


## 9 STATEMENT OF COMPLIANCE

## 9.1 Ethical and Regulatory Aspects

The clinical investigation will be carried out in accordance with the following texts:

- The Declaration of Helsinki (1996)
- Good Clinical Practice (ICH E6) (current version)
- DIN EN ISO 14155:2020

The clinical investigation will not begin until the required approval / favorable opinion from the EC and / or regulatory authority (if applicable) have been obtained. Any additional requirements imposed by the EC or regulatory authority will be followed.

Regulatory reporting responsibilities are specified in the respective Clinical Trial Agreements that also need to be duly signed prior to the first enrollment.

Quality Control and Quality Assurance systems will ensure that the clinical investigation is conducted according to local law and Good Clinical Practices. Olympus Europa SE & Co. KG will follow their own Standardized Operating Procedures covering all aspects of the clinical investigation.

## 9.2 Patient Coverage

The PowerSpiral medical device is a CE-certified and CE-marked product. Any patient product liability claims will be covered in accordance with the applicable product liability law. Additional patient coverage will be provided by the sponsor if required by national law.

#### 9.3 Retention of Documents

The investigator must conduct the study in compliance with the Medical Devices Act and Good Clinical Practices. The study documents comprise the following:

- Case report forms,
- Data correction/clarification forms,
- Source documents,
- Correspondence between sponsor/CRO and investigator,
- Regulatory documents such as:
  - Signed CIP and any amendments,
  - > EC approval and correspondence,
  - Curriculum Vitae of medical personnel (investigators, study nurses, etc.),
  - Subject signed consent forms,
  - Investigator's contract


Source documents for study subjects shall be marked with the CIP Reference number [2018-GI (OEKG) -01].

The CIP, case report forms, correspondence, original informed consent forms, subject identification log with names of the patients and other documents concerning the study must be kept by the investigator in the investigator site file according to local regulations. The safekeeping period is usually 15 years after study close-out.

## 9.4 Auditing procedures

National or foreign Health authorities may want to inspect your site at any time during or after the study. By participating in this clinical investigation investigators agree to and will grant authorized inspectors access to all original documents, including subject files. If subject files or medical records are stored on a computer system, the investigator (or delegate) shall ensure that data requested by the inspector is printed on paper, dated and signed before handed over to the inspector. Inspectors do not have direct access to the sites computer system.

Also the sponsor (Olympus Europa SE & Co. KG) reserves the right to perform an audit during the active study phase or after study closeout.


## 10 INFORMED CONSENT

Before enrolment in the clinical investigation, the investigator must make sure that all eligible subjects are well provided with detailed information, both orally and in writing, about the following points in particular:

- · Aims, duration and methods of the clinical investigation.
- Risks, anticipated benefits and potential hazards according to current knowledge.
- That he/she is free to withdraw his/her consent at any time without affecting subsequent treatment or his/her relation to the physician.
- That the clinical research monitors and auditors, Health Authority Inspectors and EC/IRB members may have access to their clinical source data.

Informed consent must be given by a standard written declaration drafted in simple non-technical language. Subjects will also be informed that the data collected during the study will be archived and processed in accordance with local individual data protection law.

The subject must read and understand the contents of this form before signing and dating it. He/she has to be provided with a signed version. No subject may be enrolled in this clinical investigation before giving his/her informed consent in writing.

The investigator will inform all subjects included in the clinical investigation about any new information on the investigational device discovered during the study, in accordance with the recommendations of Olympus Europa SE & Co. KG, the sponsor, and the EC.

The investigator must hold an updated list of all subjects enrolled in the study by recording their subject number. A Subject Identification Log Template will be provided by the sponsor.


# 11 ADVERSE EVENTS, ADVERSE DEVICE EFFECTS AND DEVICE DEFICIENCIES

## 11.1 Definitions (according to ISO 14155:2020)

#### 11.1.1 Adverse event (AE)

The term AE describes any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including laboratory values) in subjects, users or other persons, whether or not related to the investigational medical device. For subjects this definition includes:

- Events related to the investigational medical device
- Events related to the procedures involved
- For users or other persons, this definition is restricted to events related to investigational medical devices

#### Note:

A "significant deterioration in laboratory parameters" means an abnormal lab value, which is deemed clinically significant when any of the following conditions is met:

- The abnormality suggests a disease and/or organ toxicity that is new or has worsened from baseline.
- The abnormality is of a degree that requires additional active management, e.g. change of treatment, discontinuation of treatment, close observation, more frequent follow-up assessments, or further diagnostic investigation.

Therefore, a clinically significant deterioration of a lab value is one that indicates a new disease process, worsening of an existing condition, or requires further action(s) to be taken.

### 11.1.2 Adverse Device Effect (ADE)

An ADE is an adverse event related to the use of an investigational medical device.

#### Note:

- This definition includes any adverse event resulting from insufficiencies or inadequacies in the instructions for use, the deployment, the implantation, the installation, the operation, or any malfunction of the investigational medical device.
- This definition includes any event that is a result of a use error or intentional misuse.
- This includes medical devices already on the market that are being evaluated for unintended uses, new populations, new materials or design changes.


## 11.1.3 Serious Adverse Event / Serious Adverse Device Effect (SAE /SADE)

A SAE/SADE is further specified by the fact that it results or could have resulted in death or severe deterioration of health of a subject, user, or other persons, whether (SADE) or not (SAE) related to the investigational medical device.

The criteria for a Serious Adverse Event (SAE) are the following:

- Led to a death,
- Led to a serious deterioration in health of the subject, that either resulted in:
  - > A life-threatening illness or injury, or
  - A permanent impairment of a body structure or a body function, or
  - In-patient or prolonged hospitalization, or
  - > In medical or surgical intervention to prevent life threatening illness or injury or permanent impairment to a body structure or a body function,
- Led to fetal distress, fetal death or a congenital abnormality or birth defect.

**Note:** Planned hospitalization for a pre-existing condition, or a procedure required by the CIP, without serious deterioration in health, is not considered a serious adverse event.

The following points should be taken into account when evaluating the seriousness of an Adverse Event:

- The life-threatening criterion indicates that there was an immediate risk of death at the time
  of its occurrence. This does not mean that if the adverse event had occurred in a more
  severe form it would have led to death.
- The following events are not considered to be serious adverse events:
  - An event causing a brief visit to a hospital consultation, an open-door or day hospital.
  - Outpatient treatment in the emergency department although the reason for which this treatment was instituted may be serious.
  - Admission to hospital (more than one night in a hospital bed) including surgical operations planned before or during the study if the condition was present before the study and provided that it does not worsen during the study.

#### Note:

A state of pregnancy is an exclusion criterion. Hence contraceptive measures must be taken by all subjects of childbearing potential throughout the study. However, if pregnancy is discovered during the study, the study participation must be discontinued immediately and the outcome of the pregnancy must be followed up carefully. Any abnormal outcome of the child or the mother must be documented.


#### 11.1.4 Device Deficiencies

Device Deficiencies means any inadequacy of a medical device with respect to its identity, quality, durability, reliability, safety or performance

#### 11.2 Documentation

#### 11.2.1 (Serious) Adverse Events / Adverse Device Effects

Independent from a possible relation to the investigational device, every AE spontaneously reported by the subject or observed by the investigator will be reported on the appropriate page of the case report form. Furthermore, the investigator shall actively ask the subject about the occurrence of any (S)AE at each visit and note any abnormal laboratory findings. For each adverse event the following information shall be documented:

- Description of the event (diagnosis and symptoms in verbatim terms). For the most common ERCP-related adverse events the following terms could be selected:
  - Pancreatitis
  - Cholangitis
  - Cholecystitis
  - Bleeding
  - Perforation (according (Stapfer 2000)
    - Type I Duodenal wall perforation (by the endoscope)
    - Type II Periampullary perforation (by sphincterotomy/ precut)
    - Type III Biliary or pancreatic duct perforation (by intraductal instrumentation
    - Type IV Retroperitoneal gas alone
  - Sedation-related AEs
- Outcome,
- Seriousness,
- Duration (start date and stop date),
- Causal relationship to the investigational device.
   Causality assessment will be done by the investigator using a 5-category system (no related / unlikely / possible / probable / causal relationship).
- Any therapy or corrective action initiated including.

The results of any complementary tests performed (laboratory tests, ECG, etc.) must be pseudonymized by the investigator prior to forwarding information to the sponsor. A period of 4 weeks for follow up of AEs after the subject has routinely completed or prematurely terminated the study seems sufficient. This means that any additional information needed to assess the (S)AE should be collected and documented in the respective CRF within one month after occurrence.


11.2.2 **Device deficiencies** 

Two device deficiencies of the disposable Spiral Segment were documented in previous clinical

studies with PowerSpiral. The technical issues are addressed and solved.

**Reporting Responsibilities** 11.3

11.3.1 Serious Adverse Events (SAE) / Serious Adverse Device Effects (SADE)

After the signature on the consent form is obtained, any SAE occurring while the subject is enrolled

in the study must be immediately reported by the investigator.

11.3.1.1 **Serious Adverse Event - Initial Report** 

The investigator has to report every SAE immediately after he/she becomes aware of the SAE.

The Sponsor compile an accumulated SAE list and share with Ethical Committees on a bi-annual

basis (if requested by the respective Ethical Committees). However, for international safety

reporting requirements the sponsor needs to be informed immediately about any observed SAE.

11.3.1.2 Serious Adverse Event - Follow-up Report

If the event / SAE is not resolved further information (e.g. laboratory reports, surgical reports) for

full assessment is needed and shall be provided as soon as it becomes available. The sponsor

may request additional documents, shall be provided within 5 days.

11.3.2 **Device deficiencies** 

Device deficiencies shall be reported to the sponsor not later than 7 working days after observation.

11.3.3 **Responsible Nominated Safety Contact** 

Peter Teichmann, PhD

Manager Clinical Operations

OLYMPUS EUROPA SE & Co. KG

email: <a href="mailto:peter.teichmann@olympus-europa.com">peter.teichmann@olympus-europa.com</a>

phone: +49 40 23773 7835

mobile: +49 170 5570 674

fax: +49 40 23773 507835

The sponsor will monitor the safety of the PowerSpiral device in particular for the Endoscopic

Retrograde Cholangiopancreatography. All SAEs will be checked on a case-by-case basis by an

independent, external expert.


## 11.4 Anticipated Adverse Events

Foreseeable risks include those typically associated with ERCP performed under general anesthesia or sedation.

The following device and process related events were observed in previous Investigator-Initiated-Trials with PowerSpiral and reported in the context of post-market surveillance. The SAMISEN study will contribute and extend the safety profile of the PowerSpiral device.


## Table 2 List of anticipated (Serious) Adverse Events

- tissue damage
- mucosal damage
- laceration
- inflammation
- bleeding
- hematoma
- perforation
- penetration
- infection
- pain (such as abdominal pain sore throat and odynophagia)
- abdominal distention
- discomfort (such as abdominal discomfort and swallowing discomfort)
- indigestion
- nausea
- vomiting
- cardiovascular problem (bradycardia, tachycardia, hypotension and hypertension)
- dysphagia
- respiratory system disorder (such as aspiration pneumonia, cough, hypoxemia, respiratory instability and mediastinal emphysema)
- pancreatitis
- fever
- hyperamylasemia
- hyperlipasemia
- intestinal obstruction
- intestinal necrosis
- intussusception
- parotitis
- hiccup
- electrical shock
- burn (oerator)
- physical deconditioning
- distress
- allergy
- heat injury
- exposure
- acute pancreatitis
- cholangitis
- aspiration pneumonia
- CO2 narcosis
- atrioventricular block
- surgery (as a result of perforation, laceration, bleeding, tissue damage, etc)
- bruise (Health Care Professional)
- bleeding (Health Care Professional)


# 11.5 Data Monitoring Committee

Not applicable.


# 12 VULNERABLE POPULATION

It is not planned to include a vulnerable population.


# 13 SUSPENSION OR PREMATURE TERMINATION

Certain circumstances may lead to early termination of an entire clinical investigation, in particular for ethical or safety reasons such as:

- The high frequency and/or unexpected severity of adverse events.
- Unsatisfactory recruitment of subjects as far as their quantity or quality is concerned or recurrent incomplete/inappropriate collection of data.

The decision to put a study on hold or for premature termination will be made by the Sponsor.


## 14 PUBLICATION POLICY

The sponsor is explicitly committed to publish the trial results in a scientific medical journal and / or presented at scientific meetings. The Investigator agrees that any publication by the Study Site of study results conducted at their study site shall not be made before the first multicenter publication and as agreed between the sponsor and the Coordinating Clinical Investigator.

For greater certainty, it is hereby recalled that in its capacity as sponsor of the trial, Olympus Europa SE & Co. KG is solely responsible to co-ordinate the publications of multicenter clinical trials in order to ensure that the related results are reported in a coherent and responsible manner so that results from clinical trial data subsets are not published in advance of or without clear reference to the primary publication and/or do not repeat such primary publication. Olympus Europa SE & Co. KG decides about the nomination of investigators as authors on the basis of its internal policies, requirements of the publishers and generally accepted standards of authorship. Therefore, Olympus Europa SE & Co. KG shall be duly informed of any publication plans in order to review any proposed manuscript before submission for publication.


## 15 BIBLIOGRAPHY

- Akarsu, M., S. Akkaya Ozdinc, A. Celtik, and H. Akpinar. 2014. 'Diagnostic and therapeutic efficacy of double-balloon endoscopy in patients with small intestinal diseases: single-center experience in 513 procedures', *Turk J Gastroenterol*, 25: 374-80.
- Akerman, Paul A., and Daniel Cantero. 2009. 'Severe Complications of Spiral Enteroscopy in the First 1750 Patients', *Gastrointestinal Endoscopy*, 69.
- Aktas, H., L. de Ridder, J. Haringsma, E. J. Kuipers, and P. B. Mensink. 2010. 'Complications of single-balloon enteroscopy: a prospective evaluation of 166 procedures', *Endoscopy*, 42: 365-8.
- Anvari, S., Y. Lee, N. Patro, M. S. Soon, A. G. Doumouras, and D. Hong. 2021. 'Double-balloon enteroscopy for diagnostic and therapeutic ERCP in patients with surgically altered gastrointestinal anatomy: a systematic review and meta-analysis', *Surg Endosc*, 35: 18-36.
- Arulanandan, A., P. S. Dulai, S. Singh, W. J. Sandborn, and D. Kalmaz. 2016. 'Systematic review: Safety of balloon assisted enteroscopy in Crohn's disease', *World J Gastroenterol*, 22: 8999-9011.
- Beyna, T., M. Arvanitakis, M. Schneider, C. Gerges, D. Boing, J. Deviere, and H. Neuhaus. 2020. 'Motorised spiral enteroscopy: first prospective clinical feasibility study', *Gut*.
- Beyna, T., M. Arvanitakis, M. Schneider, C. Gerges, J. Hoellerich, J. Deviere, and H. Neuhaus. 2020. "Total motorized spiral enteroscopy: first prospective clinical feasibility trial." In *Gastrointest Endosc*.
- Beyna, Torsten, Markus Schneider, Jörg Höllerich, and Horst Neuhaus. 2020. "Motorized spiral enteroscopy—assisted ERCP after Roux-en-Y reconstructive surgery and bilioenteric anastomosis: first clinical case." In *VideoGIE*, 311-13.
- Dumonceau, J. M., C. Kapral, L. Aabakken, I. S. Papanikolaou, A. Tringali, G. Vanbiervliet, T. Beyna, M. Dinis-Ribeiro, I. Hritz, A. Mariani, G. Paspatis, F. Radaelli, S. Lakhtakia, A. M. Veitch, and J. E. van Hooft. 2020. "ERCP-related adverse events: European Society of Gastrointestinal Endoscopy (ESGE) Guideline." In *Endoscopy*, 127-49.
- He, Q., Y. Bai, F. C. Zhi, W. Gong, H. X. Gu, Z. M. Xu, J. Q. Cai, D. S. Pan, and B. Jiang. 2013. 'Double-balloon enteroscopy for mesenchymal tumors of small bowel: nine years' experience', *World J Gastroenterol*, 19: 1820-6.
- Krutsri, C., M. Kida, H. Yamauchi, T. Iwai, H. Imaizumi, and W. Koizumi. 2019. 'Current status of endoscopic retrograde cholangiopancreatography in patients with surgically altered anatomy', *World J Gastroenterol*, 25: 3313-33.
- Lennon, A. M., S. Kapoor, M. Khashab, E. Corless, S. Amateau, K. Dunbar, V. Chandrasekhara, V. Singh, and P. I. Okolo, 3rd. 2012. 'Spiral assisted ERCP is equivalent to single balloon assisted ERCP in patients with Roux-en-Y anatomy', *Dig Dis Sci*, 57: 1391-8.
- M Schneider, H Neuhaus, T Beyna. 2020. 'Motorized Spiral Enteroscopy-Assisted ERCP in Altered Gastrointestinal Anatomy: First Clinical Series', *United European Gastroenterol J*, 8: 144-887.
- Mans, L., M. Arvanitakis, H. Neuhaus, and J. Deviere. 2018. 'Motorized Spiral Enteroscopy for Occult Bleeding', *Dig Dis*, 36: 325-27.
- Moeschler, O., and M. K. Mueller. 2015. 'Deep enteroscopy indications, diagnostic yield and complications', *World J Gastroenterol*, 21: 1385-93.
- Moreels, T. G. 2019. 'Endoscopic retrograde cholangiopancreatography in roux-en-Y gastric bypass patients', *EDIZIONI Minerva MeDiCa*.
- Neuhaus, H., T. Beyna, M. Schneider, and J. Deviere. 2016. 'Novel motorized spiral enteroscopy: first clinical case', *VideoGIE*, 1: 32-33.
- Rondonotti, E., C. Spada, S. Adler, A. May, E. J. Despott, A. Koulaouzidis, S. Panter, D. Domagk, I. Fernandez-Urien, G. Rahmi, M. E. Riccioni, J. E. van Hooft, C. Hassan, and M. Pennazio. 2018. 'Small-bowel capsule endoscopy and device-assisted enteroscopy for diagnosis and treatment of small-bowel disorders: European Society of Gastrointestinal Endoscopy (ESGE) Technical Review', *Endoscopy*, 50: 423-46.
- Shah, R. J., M. Smolkin, R. Yen, A. Ross, R. A. Kozarek, D. A. Howell, G. Bakis, S. S. Jonnalagadda, A. A. Al-Lehibi, A. Hardy, D. R. Morgan, A. Sethi, P. D. Stevens, P. A. Akerman, S. J. Thakkar, and B. C. Brauer. 2013. 'A multicenter, U.S. experience of single-balloon, double-balloon, and


- rotational overtube-assisted enteroscopy ERCP in patients with surgically altered pancreaticobiliary anatomy (with video)', *Gastrointest Endosc*, 77: 593-600.
- Skinner, M., D. Popa, H. Neumann, C. M. Wilcox, and K. Monkemuller. 2014. 'ERCP with the overtube-assisted enteroscopy technique: a systematic review', *Endoscopy*, 46: 560-72.
- Stapfer, M., Selby, R. R., Stain, S. C., Katkhouda, N., Parekh, D., Jabbour, N., Garry, D. 2000. 'Management of duodenal perforation after endoscopic retrograde cholangiopancreatography and sphincterotomy', *Ann Surg*.


# **16 STUDY TIMELINE**

| Screening period | November 2021 – December 2022 |
|-----------------------|-------------------------------|
| Recruitment period: | November 2021 – December 2022 |
| Database lock | February 2023 |
| Data Review Meeting | February 2023 |
| Statistical analysis: | April 2023 |
| First data available | May 2023 |
| Draft report: | August 2023 |
| Final CIR | September 2023 |


## 17 ANNEX 01: DEEP ENTEROSCOPY PROCEDURE

#### 17.1 General Information

A lack of frequent stalling of the rotation should be interpretive as a warning to assess the patient and scope position.

Continued rotation without advancement should also be seen as maximum insertion depth.

The limit function does not guarantee the safety of the procedure. The operator must judge if safe insertion can be continued on a case-by-case basis.

#### The LIMIT Function?

The limit function stops the rotation of the single use PowerSpiral tube when the electric current to the motor on the endoscope a setting value. To release, remove your foot from the pedal on foot switch.

## 17.2 General Insertion tips

Gentle forward pressure is used when rotation is started as well as throughout the procedure.

Minimal CO<sub>2</sub> insufflation is recommended as small bowel distention will decrease spiral advancement.

Irrigation using a water jet may help with lumen visualization and spiral advancement Intermittent external abdominal compression is often helpful to facilitate engagement and advancement of the spiral segment.

### 17.3 General Withdrawal tips

Insufflation may be used at will at this time.

Although the scope may seem to be moving out of the patient quickly, it is important to keep holding the scope firmly.

Slow controlled withdrawal is the key. This is accomplished by backward rotation while maintaining the scope position and keeping the tip in motion


## 17.4 Antegrade Approach

## 17.4.1 Inserting the Scope

After passage of the bougie, the tip of the scope is advanced through the mouthpiece into proximal esophagus.



Rotation is started when the spiral segment is in the proximal pharynx. Begin with slow rotation with gentle pressure if needed, and the esophagus is intubated under direct visualization.



#### Note

If significant resistance is encountered during esophageal intubation, the endoscope should be removed and the esophagus should be assessed.

If no stricture is observed or motor stalls frequently, consider passage of a large bougie dilator (54-60 Fr) prior to reintroduction of the PowerSpiral.

A second attempt may be tried, with deflation of endotracheal balloon considered, but if stalling continues the procedure image is generated is smaller in caliber than the rotary


## 17.4.2 Passing through the Pharynx & Esophagus

The spiral segment is engaged in the upper esophageal sphincter and rotational advancement is continued using the forward foot switch.



The patient's neck is extended as needed to straighten the passage through the cervical esophagus as the rotating spiral section is less flexible than the remaining section of the scope.



Once the spiral section is past the cervical esophagus, the patient's neck no longer needs to be extended and may be returned to the usual position



#### Note

Gentle forward pressure is applied while the spiral segment is rotated slowly and intermittently using the foot switch facilitating intubation of the esophagus.

A decrease in the amount of resistance and torque required for advancement is an indicator that the cervical esophagus has been passed.


## 17.4.3 Passing through the Stomach

Upon entering the stomach, gastric contents should be aspirated and CO<sub>2</sub> insufflation should be kept to minimum.



While on the stomach, gentle pushing with rotation of the spiral segment is recommended for advancement.



When the insertion tube mark at 80cm is in the mouthpiece, the entire spiral segment is in the stomach.




## 17.4.4 Passing through the Duodenum

The duodenum and proximal jejunum are fixed. Passage through the segment is accomplished with forward rotation and gentle advancement of the scope.



Avoid prolonged rotation when the spiral segment is in the second portion of the duodenum.



Looping should be avoided but can be managed careful withdrawal of the scope along with forward rotation of the spiral segment.



Fluoroscopy or ScopeGuide may be useful in assessing looping.


## 17.4.5 Passing through the Small Bowel Distal to the Ligament of Treitz

Once the spiral segment is positioned in the proximal jejunum, advancement is accomplished primarily by rotation of the spiral segment.



Intermittent gentle advancement of the scope in 3-5cm increments when progress seems to slow down visually.



Insert as if drawing concentric circles.




## 17.4.6 Reaching the Terminal Ileum

The following images will provide indication of the scope being close to the terminal illeum.

The ileum becomes apparent with less prominent villi and prominent lymphoid follicles.



The procedure should be terminated if the cecum is encountered.



Do not pass the spiral through the ileo-cecal valve. Stop forward advancement.




## 17.4.7 Withdrawal Techniques

Gentle forward pressure should be maintained to facilitate a slow, controlled withdrawal. This is especially true when the duodenum is encountered.



Every effort should be made to be sure the spiral segment is free in the stomach and no longer engaged in the duodenum/ pylorus prior to allowing the spiral segment to engage the lower esophagus sphincter. This is often accomplished by intermittent use of the forward foot switch to confirm disengagement in the stomach. tent use of the forward foot switch to confirm disengagement in the stomach.



The PowerSpiral enteroscope has a special marking at 80cm to indicate the spiral segment is approaching the lower esophagus sphincter.




As the spiral segment encounters the cervical esophagus, the neck is once again extended to facilitate atraumatic withdrawal while the spiral segment is rotating.



#### Note

Increased resistance is an indicator of remaining pleated bowel on the spiral segment. This requires advancement of the scope holding position and then resuming backward rotation.


# 17.5 Retrograde Approach

### 17.5.1 Passing through the Colon

The spiral enteroscope can be passed through the colon with continuous rotation and gentle pressure.



Forward rotation of the spiral segment should be used for passage through the anal sphincter.



If lumen cannot be visualized, rotate with caution to advance.

CO₂ insufflation should be minimized and water injection should be considered.


# 17.5.2 Eliminating a Loop

Eliminate a loop by maintaining position of the spiral segment and withdrawing the scope while applying forward rotation to the spiral segment.

Sigmoid Colon:








### Transverse Colon:











## Tips

The principal is to minimize the amount of scope inserted in the colon thereby preserving as much scope length as possible with which to examine the small bowel. This is accomplished by minimizing insufflation, and the constant use of withdrawing, torquing, shortening, and pleating techniques.


## 17.5.3 Passing through the Ileo-cecal Valve

The ileocecal valve is intubated using standard colonoscopy techniques.



When passing through the ileocecal valve, insertion can be facilitated by decreasing the angle of insertion into the ileum by means of manual compression or postural change.



If insertion into the terminal ileum is still difficult, try retro-flexing the scope inside the cecum and inserting the U-shaped distal end of the scope into the ileum with a push-pull technique.

After passing through the ileocecal valve, advancement is accomplished by rotation of the spiral segment and intermittent advancement of the scope through the rectum as well as intermittent manual compression to facilitate acquisition of the small bowel on to the insertion tube.




## 17.5.4 Passing through the Small Bowel

Once the spiral segment is positioned in the terminal ileum, advancement is accomplished primarily by rotation of the spiral segment and intermittent gentle advancement of the scope in 3-5 cm increments when progress seems to slow down visually.



## 17.5.5 Reaching the Proximal Jejunum

The following images will provide indication of the scope being close to the proximal jejunum.

The procedure should be terminated if the ampulla or duodenal bulb is encountered.




## 17.5.6 Withdrawal Techniques

Slow withdrawal is accomplished with the foot switch in the reverse position and constant maneuvering of the scope tip to facilitate gradual and controlled release of the intestine off the tip of the scope.



Occasional forward activation of the spiral may be necessary for a slow, controlled withdrawal.



Once the cecum is reached, the scope is withdrawn as in a standardized colonoscopy with or without spiral rotation.




When the anal sphincter is reached, the passage is accomplished by the spiral rotation in the backward direction.



## Note

Retroflextion should not be performed with the spiral segment in the patient.